CLINICAL TRIAL: NCT00348751
Title: The Effect of Alerting Versus on Demand Computer Based Decision Support on Treatment of Dyslipidaemia by General Practitioners - The CholGate Randomized Trial
Brief Title: CholGate - The Effect of Alerting Versus on Demand Computer Based Decision Support on Treatment of Dyslipidaemia by General Practitioners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2000B161
Record Dates: First submitted 2006-06-29; First posted 2006-07-06 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2006-06

CONDITIONS: Decision Support Systems, Clinical

INTERVENTIONS:
Device: CholGate

SUMMARY:
Indirect evidence show alerting physicians with clinical decision support systems (CDSS) seem to change behaviour more than requiring users to actively initiate the system. However, randomized trials comparing these methods in a clinical setting are lacking. In this study we compare the effect of Alerting physicians with a CDSS or actively requiring initiation of CDSS on the adherence of Dutch general practitioners to the Cholesterol guideline of the Dutch college of General Practitioners.

DETAILED DESCRIPTION:
Indirect evidence show alerting physicians with clinical decision support systems (CDSS) seem to change behaviour more than requiring users to actively initiate the system. However, randomized trials comparing these methods in a clinical setting are lacking. In this study we compare the effect of Alerting physicians with a CDSS or actively requiring initiation of CDSS on the adherence of Dutch general practitioners to the Cholesterol guideline of the Dutch college of General Practitioners, using a clinical decsion support system called CholGate. This system has the functionality to provide both Alerting and On-Demand decision support. Users are free to negate the advise provided by the decision support system. The trial will have a cluster randomized structure.

ELIGIBILITY:
Inclusion Criteria:

* All general practices using only Elias electronic patient records (ISOFT b.V)
* All patients meeting the screening and treatment criteria of the Dutch college of general practitioners cholesterol guideline

Exclusion Criteria:

* Practices that used paper based records

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Study Completion 2005-11

PRIMARY OUTCOMES:
The percentage of correctly screened patients using anonymous patient record data.
The percentage of correctly treated patients using anonymous patient record data.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus T van Wyk, MD, PhD, Principal Investigator — ErasmusMC University Medical Centre Rotterdam
Locations (1):
- Department of Medical informatics, ErasmusMC, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Van Wyk JT, Van Wijk MA, Moorman PW, Mosseveld M, Van Der Lei J. Cholgate - a randomized controlled trial comparing the effect of automated and on-demand decision support on the management of cardiovascular disease factors in primary care. AMIA Annu Symp Proc. 2003;2003:1040. PMID 14728543
- [Background] Van Wyk JT, Van Wijk MA. Assessment of the possibility to classify patients according to cholesterol guideline screening criteria using routinely recorded electronic patient record data. Stud Health Technol Inform. 2002;93:39-46. PMID 15058412
- [Background] Van Wyk JT, Van Wijk MA. Analysis of Dutch general practice guidelines for inconsistencies with respect to the management of cardiovascular disease risk factors. Stud Health Technol Inform. 2004;107(Pt 1):179-86. PMID 15360799
- [Background] van Wyk JT, Picelli G, Dieleman JP, Mozaffari E, Kramarz P, van Wijk MA, van der Lei J, Sturkenboom MC. Management of hypertension and hypercholesterolaemia in primary care in The Netherlands. Curr Med Res Opin. 2005 Jun;21(6):839-48. doi: 10.1185/030079905X46368. PMID 15969884
- [Background] Dieleman JP, van Wyk JT, van Wijk MA, van Herpen G, Straus SM, Dunselman H, Sturkenboom MC. Differences between statins on clinical endpoints: a population-based cohort study. Curr Med Res Opin. 2005 Sep;21(9):1461-8. doi: 10.1185/030079905X61866. PMID 16197665
- [Background] van Wyk JT, van Wijk MA, Sturkenboom MC, Moorman PW, van der Lei J. Identification of the four conventional cardiovascular disease risk factors by Dutch general practitioners. Chest. 2005 Oct;128(4):2521-7. doi: 10.1378/chest.128.4.2521. PMID 16236918
- [Background] van Wyk JT, van Wijk MA, Moorman PW, van der Lei J. Cross-sectional analysis of guidelines on cardiovascular disease risk factors: going to meet the inconsistencies. Med Decis Making. 2006 Jan-Feb;26(1):57-62. doi: 10.1177/0272989X05284104. PMID 16495201
- [Background] van Wyk JT, van Wijk MA, Moorman PW, Mosseveld M, van der Lei J. User requirements rating and knowledge-level of general practitioners at the start of CholGate - a lipid management decision support project. AMIA Annu Symp Proc. 2005;2005:1146. PMID 16779432